CLINICAL TRIAL: NCT06274918
Title: Reducing Intraoperative ESKAPE (Enterococcus, S. Aureus, Klebsiella, Acinetobacter, Pseudomonas, and Enterobacter Spp.) Transmission Via Use of an Evidence-Based, Hand Hygiene Program Optimized by OR PathTrac
Brief Title: Reducing ESKAPE Transmission in the Operating Room
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: RDB Bioinformatics (Industry); Georgia-Pacific (Unknown)
Responsible Party: Principal Investigator, Andrew Pugely, Principle Investigator, University of Iowa
Other Study IDs: 202111418
Record Dates: First submitted 2023-01-31; First posted 2024-02-23 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Surgical Procedure, Unspecified

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples With DNA — We will be collecting bacterial pathogens from anesthesia work area reservoirs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Usual care: Patients undergoing surgery requiring general anesthesia. Usual hand hygiene devices and products will be accessible which will include but are not limited to those mounted to the wall outside of the operating room entrance and those present on the anesthesia cart.
- Personalized body worn alcohol dispenser: Anesthesia providers (attending anesthesiologist and their assistant (resident physician/Certified-Registered Nurse Anesthetist (CRNA), or student nurse assistant (SRNA) will receive a personalized, body worn alcohol dispenser in addition to usual hand hygiene devices/products for hand decontamination during surgery requiring general anesthesia.
  Interventions: Device: Personalized Body-Worn Alcohol Dispenser

INTERVENTIONS:
Device: Personalized Body-Worn Alcohol Dispenser — This is an alcohol dispenser that will be worn on the Anesthesia Providers scrub pants, near the hip. It will be worn by both the attending physician and the resident physician/CRNA/SRNA. The device is produced by Georgia-Pacific.
  Groups: Personalized body worn alcohol dispenser

SUMMARY:
This study is designed to examine the impact of a personalized, body worn alcohol dispenser on the epidemiology of ESKAPE transmission in the anesthesia work area for patients undergoing surgery requiring general anesthesia.

DETAILED DESCRIPTION:
A solid body of published and preliminary evidence leveraging systematic phenotypic and whole cell genome analysis and innovative surveillance technology has provided great insight into the epidemiology of perioperative bacterial transmission and healthcare-associated infection (HAI) development. This work has led us to three primary assertions that serve as the foundation of our scientific premise: 1) Further progress towards HAI prevention is needed, 2) Prevention of perioperative ESKAPE transmission is an important improvement target, and 3) An evidence-based, multi-faceted program can reduce perioperative ESKAPE transmission. Further work to generate intraoperative hand hygiene improvement is indicated. We hypothesize that the proposed program will generate sustained reductions in OR ESKAPE exposure and S. aureus transmission that will lead to sustained reductions in perioperative HAIs.

ELIGIBILITY:
Inclusion Criteria: Adult patients undergoing surgery requiring general anesthesia and peripheral IV and/or central line placement.

Exclusion Criteria:

Pediatric patient, not requiring general anesthesia and/or IV/central line placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing surgery requiring general anesthesia and intravascular access.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
ESKAPE transmission events with and without the body worn device | Up to 96 hours from the surgial procedure
  Reduce the number of Enterococcus, Staphylococcus aureus, Pseudomonas, and other gram-negative (i.e., Klebsiella, Acinetobacter, Pseudomonas, and Enterobacter spp.) transmission events

SECONDARY OUTCOMES:
The epidemiology of ESKAPE transmission events | Up to 90 days from surgery
  To characterize the epidemiology of ESKAPE transmission with and without the device according to incidence.
The epidemiology of ESKAPE transmission events | Up to 90 days from surgery
  To characterize the epidemiology of ESKAPE transmission with and without the device according to reservoir of origin.
The epidemiology of ESKAPE transmission events | Up to 90 days from surgery
  To characterize the epidemiology of ESKAPE transmission with and without the device according to transmission location(s).
The epidemiology of ESKAPE transmission events | Up to 90 days from surgery
  To characterize the epidemiology of ESKAPE transmission with and without the device according to portal of entry (stopcock).
The epidemiology of ESKAPE transmission events | Up to 90 days from surgery
  To characterize the epidemiology of ESKAPE transmission with and without the device according to mode (within or between-case).
90-Day Healthcare-Associated Infections | 90 days following surgery
  Number of infections occurring within 90 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pugely, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data requests submitted to the PI will be reviewed and considered.
Supporting Information: Study Protocol
Time Frame: 1 year from the final study completion date (earliest date) and up to an additional 24 months.
Access Criteria: A sumitted proposal that is reviewed and approved by the PI

REFERENCES:
- [Background] Vogel TR, Dombrovskiy VY, Lowry SF. Impact of infectious complications after elective surgery on hospital readmission and late deaths in the U.S. Medicare population. Surg Infect (Larchmt). 2012 Oct;13(5):307-11. doi: 10.1089/sur.2012.116. Epub 2012 Oct 19. PMID 23082877
- [Background] Awad SS. Adherence to surgical care improvement project measures and post-operative surgical site infections. Surg Infect (Larchmt). 2012 Aug;13(4):234-7. doi: 10.1089/sur.2012.131. Epub 2012 Aug 22. PMID 22913334
- [Background] Kirkland KB, Briggs JP, Trivette SL, Wilkinson WE, Sexton DJ. The impact of surgical-site infections in the 1990s: attributable mortality, excess length of hospitalization, and extra costs. Infect Control Hosp Epidemiol. 1999 Nov;20(11):725-30. doi: 10.1086/501572. PMID 10580621
- [Background] Magill SS, O'Leary E, Janelle SJ, Thompson DL, Dumyati G, Nadle J, Wilson LE, Kainer MA, Lynfield R, Greissman S, Ray SM, Beldavs Z, Gross C, Bamberg W, Sievers M, Concannon C, Buhr N, Warnke L, Maloney M, Ocampo V, Brooks J, Oyewumi T, Sharmin S, Richards K, Rainbow J, Samper M, Hancock EB, Leaptrot D, Scalise E, Badrun F, Phelps R, Edwards JR; Emerging Infections Program Hospital Prevalence Survey Team. Changes in Prevalence of Health Care-Associated Infections in U.S. Hospitals. N Engl J Med. 2018 Nov 1;379(18):1732-1744. doi: 10.1056/NEJMoa1801550. PMID 30380384
- [Background] World Health Organization. Antimicrobial Resistance. Global Report on Surveillance. WHO. 2014
- [Background] German RR, Lee LM, Horan JM, Milstein RL, Pertowski CA, Waller MN; Guidelines Working Group Centers for Disease Control and Prevention (CDC). Updated guidelines for evaluating public health surveillance systems: recommendations from the Guidelines Working Group. MMWR Recomm Rep. 2001 Jul 27;50(RR-13):1-35; quiz CE1-7. PMID 18634202
- [Background] Boucher HW, Talbot GH, Bradley JS, Edwards JE, Gilbert D, Rice LB, Scheld M, Spellberg B, Bartlett J. Bad bugs, no drugs: no ESKAPE! An update from the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jan 1;48(1):1-12. doi: 10.1086/595011. PMID 19035777
- [Background] Loftus RW, Koff MD, Brown JR, Patel HM, Jensen JT, Reddy S, Ruoff KL, Heard SO, Yeager MP, Dodds TM. The epidemiology of Staphylococcus aureus transmission in the anesthesia work area. Anesth Analg. 2015 Apr;120(4):807-18. doi: 10.1213/ANE.0b013e3182a8c16a. PMID 24937345
- [Background] Loftus RW, Dexter F, Robinson ADM. High-risk Staphylococcus aureus transmission in the operating room: A call for widespread improvements in perioperative hand hygiene and patient decolonization practices. Am J Infect Control. 2018 Oct;46(10):1134-1141. doi: 10.1016/j.ajic.2018.04.211. Epub 2018 Jun 12. PMID 29907449
- [Background] Loftus RW, Dexter F, Robinson ADM. Methicillin-resistant Staphylococcus aureus has greater risk of transmission in the operating room than methicillin-sensitive S aureus. Am J Infect Control. 2018 May;46(5):520-525. doi: 10.1016/j.ajic.2017.11.002. Epub 2018 Jan 4. PMID 29307750
- [Background] Loftus RW, Dexter F, Robinson ADM, Horswill AR. Desiccation tolerance is associated with Staphylococcus aureus hypertransmissibility, resistance and infection development in the operating room. J Hosp Infect. 2018 Nov;100(3):299-308. doi: 10.1016/j.jhin.2018.06.020. Epub 2018 Jun 30. PMID 29966756
- [Background] von Eiff C, Becker K, Machka K, Stammer H, Peters G. Nasal carriage as a source of Staphylococcus aureus bacteremia. Study Group. N Engl J Med. 2001 Jan 4;344(1):11-6. doi: 10.1056/NEJM200101043440102. PMID 11136954
- [Background] Hadder B, Patel HM, Loftus RW. Dynamics of intraoperative Klebsiella, Acinetobacter, Pseudomonas, and Enterobacter transmission. Am J Infect Control. 2018 May;46(5):526-532. doi: 10.1016/j.ajic.2017.10.018. Epub 2018 Feb 12. PMID 29395508
- [Background] Loftus RW, Koff MD, Burchman CC, Schwartzman JD, Thorum V, Read ME, Wood TA, Beach ML. Transmission of pathogenic bacterial organisms in the anesthesia work area. Anesthesiology. 2008 Sep;109(3):399-407. doi: 10.1097/ALN.0b013e318182c855. PMID 18719437
- [Background] Rowlands J, Yeager MP, Beach M, Patel HM, Huysman BC, Loftus RW. Video observation to map hand contact and bacterial transmission in operating rooms. Am J Infect Control. 2014 Jul;42(7):698-701. doi: 10.1016/j.ajic.2014.02.021. PMID 24969122
- [Background] Koff MD, Loftus RW, Burchman CC, Schwartzman JD, Read ME, Henry ES, Beach ML. Reduction in intraoperative bacterial contamination of peripheral intravenous tubing through the use of a novel device. Anesthesiology. 2009 May;110(5):978-85. doi: 10.1097/ALN.0b013e3181a06ec3. PMID 19352154
- [Background] Loftus RW, Muffly MK, Brown JR, Beach ML, Koff MD, Corwin HL, Surgenor SD, Kirkland KB, Yeager MP. Hand contamination of anesthesia providers is an important risk factor for intraoperative bacterial transmission. Anesth Analg. 2011 Jan;112(1):98-105. doi: 10.1213/ANE.0b013e3181e7ce18. Epub 2010 Aug 4. PMID 20686007
- [Background] Loftus RW, Brown JR, Koff MD, Reddy S, Heard SO, Patel HM, Fernandez PG, Beach ML, Corwin HL, Jensen JT, Kispert D, Huysman B, Dodds TM, Ruoff KL, Yeager MP. Multiple reservoirs contribute to intraoperative bacterial transmission. Anesth Analg. 2012 Jun;114(6):1236-48. doi: 10.1213/ANE.0b013e31824970a2. Epub 2012 Mar 30. PMID 22467892
- [Background] Loftus RW, Patel HM, Huysman BC, Kispert DP, Koff MD, Gallagher JD, Jensen JT, Rowlands J, Reddy S, Dodds TM, Yeager MP, Ruoff KL, Surgenor SD, Brown JR. Prevention of intravenous bacterial injection from health care provider hands: the importance of catheter design and handling. Anesth Analg. 2012 Nov;115(5):1109-19. doi: 10.1213/ANE.0b013e31826a1016. Epub 2012 Oct 9. PMID 23051883
- [Background] Loftus RW, Brindeiro BS, Kispert DP, Patel HM, Koff MD, Jensen JT, Dodds TM, Yeager MP, Ruoff KL, Gallagher JD, Beach ML, Brown JR. Reduction in intraoperative bacterial contamination of peripheral intravenous tubing through the use of a passive catheter care system. Anesth Analg. 2012 Dec;115(6):1315-23. doi: 10.1213/ANE.0b013e31826d2aa4. Epub 2012 Nov 9. PMID 23144441
- [Background] Clark C, Taenzer A, Charette K, Whitty M. Decreasing contamination of the anesthesia environment. Am J Infect Control. 2014 Nov;42(11):1223-5. doi: 10.1016/j.ajic.2014.07.016. Epub 2014 Oct 30. PMID 25444268
- [Background] Sundara R. Microbial Contamination of Today's Operating Room Environments. IARS Poster Session 1431. April 29th, Hyatt Regency Chicago Hotel, Chicago, Il. Accessed June 19th, 2018.
- [Background] Dancer SJ, Stewart M, Coulombe C, Gregori A, Virdi M. Surgical site infections linked to contaminated surgical instruments. J Hosp Infect. 2012 Aug;81(4):231-8. doi: 10.1016/j.jhin.2012.04.023. Epub 2012 Jun 15. PMID 22704634
- [Background] Koff MD, Loftus RW, Burchman CA, Hogan DA, Beach ML. Microbial Contamination in the Anesthesia Workspace. Are We as Clean as We Think? Anesthesiology 2007; 107: A1788